CLINICAL TRIAL: NCT03935529
Title: Behavioural Activation for Low Mood in Multiple Sclerosis
Acronym: BALMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 181001
Record Dates: First submitted 2019-04-16; First posted 2019-05-02 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-05

CONDITIONS: Depression; Secondary-progressive Multiple Sclerosis
MeSH Terms: conditions — Depression; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Intervention Model Description: Multiple Single Case Experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioural Acitivation (Experimental): Behavioural Activation. Originally a component of cognitive behavioural therapy, Behavioural Activation is a structured psychotherapeutic approach which aims to (a) increase engagement in activities associated with pleasure or mastery, (b) decrease engagement in activities that maintain depression, and (c) problem solve barriers limiting access to reward or maintain aversive control. Behavioural Activation involves the use of activities to improve life situations or depressed mood.
  Interventions: Behavioral: Behavioural Activation

INTERVENTIONS:
Behavioral: Behavioural Activation — Participants will receive five sessions of Behavioural Activation. Behavioural Activation uses strategies such as activity scheduling, mastery and pleasure ratings, and graded task assignments to change a participant's perception of specific situations.
  Behavioural Activation is based on the behavioural model of depression (Lewinsohn & Shaffer, 1971). Specifically, that depression is a result of reduced positive reinforcement, particularly in social relationships. Behavioural Activation aims to reduce depressive symptoms by implementing a schedule of positive reinforcement by altering a participant's behaviour and/or their environment. As, in certain environmental contexts, behaviours that reduce depression will continue to occur through reinforcement and those that increase depression will decrease over time (Roane, Fisher, & Carr, 2016).
  Behavioural Activation has been shown to be an effective intervention for the reduction of depressed mood.

SUMMARY:
Title: Behavioural Activation for Low mood in Multiple Sclerosis The study will be sponsored by the University of Lincoln, indemnity will be provided by U M Association Limited.

Depression is highly prevalent among people with Multiple Sclerosis (MS). More specifically, as the disease progresses, people are more likely to develop depression and there is limited evidence of suitable interventions in this group. There are few studies that investigate the most appropriate duration, delivery modality, or individual adaptations for therapy for people with secondary progressive Multiple Sclerosis. This is problematic because continued reduction in physical and cognitive ability, combined with greater incidence of depression, may make accessing and engaging in therapies difficult.

Behavioural activation is a technique used as a component of psychotherapy. Behavioural activation aims to reduce behaviours that maintain or exacerbate depression by promoting counteracting behaviours, using strategies such as activity monitoring and scheduling.

However, there is no research looking in-depth at the underlying processes. Therefore, this research aims to explore the feasibility and efficacy of behavioural activation by:

* Adapting an existing behavioural activation manual into five sessions, suitable for people with secondary progressive MS.
* Examining if behavioural activation is followed by phases of change that are considered to predict later therapeutic outcome and to determine whether behavioural activation accounts for changes observed.

Up to ten participants from Nottingham University Hospitals will be recruited. Participants will be briefed on the research aims and consent will be obtained before commencing the intervention. The project will follow a multiple baseline single-case experimental design. Participants will complete weekly outcome measures that aim to observe low mood, quality of life, and adherence to behavioural activation and alignment with individual's values. Following five to six contact sessions, participants will take part in a follow-up interview. Participants will then be debriefed.

DETAILED DESCRIPTION:
The study aims will be achieved using a single centre, mixed-methods design, over two phases. The first phase will be the adaptation of an existing behavioural activation manual. The aims of the second phase will be achieved using a multiple single-case experimental design and change interview. The multiple single-case experimental design will use an AB design where each participant is their own control.

Participants will be recruited from the Nottingham University Hospitals Trust by the multiple sclerosis (MS) clinical care team, who will provide participants with the study advertisement. The initial approach will be from a member of the patient's usual care team (which may include the investigator), and information about the trial will be on display in the relevant areas. Participants can also self-refer, using information from study-related advertisements placed in the MS clinics, MS Society local branch newsletters and social media. The study aims to recruit up to ten participants. A convenience sampling technique will be used to recruit participants. Following the identification of potential participants, the intervention will be conducted by telephone, internet video-calling software, and face-to-face meetings at the participant's home.

The investigator or their nominee, e.g. from the research team or a member of the participant's usual care team, will inform the participant or their nominated representative (other individual or other body with appropriate jurisdiction), of all aspects pertaining to participation in the study.

Participants will receive a screening and information pack, containing a consent form, participant information sheet, and Hospital Anxiety and Depression Scale. A telephone call from the researcher will provide opportunity for further questions. If the participant does not meet the inclusion criterion, they will be excluded and provided with an information sheet for managing emotions.

It will be explained to the potential participant that entry into the trial is entirely voluntary and that their treatment and care will not be affected by their decision. It will also be explained that they can withdraw at any time, but attempts will be made to avoid this occurrence. In the event of their withdrawal it will be explained that their data collected so far may not be erased in accordance with the University's Research Privacy Notice and information given in the Participant Information Sheet and the investigators will seek consent to use the data in the final analyses where appropriate.

Following the interview, participants will be thanked for their time with a £20 Amazon voucher.

Study as experienced by the participant:

Following recruitment, participants will be sent instructions for installing video communication software (e.g., Skype). The researcher will contact the participant to complete pre-intervention measures and collect demographic and clinical information. Following the contact, participants will complete the baseline measure every-other-day to establish a baseline. Participants will complete measures using Qualtrics (a data management service).

A baseline will be established over two weeks for each participant in which no other contact or procedure will be introduced. The baseline will be considered stable (established) when the participant has recorded no less than three data points on the baseline measure that show no trend toward improvement. If stability has not been demonstrated, the baseline will be extended on a week-by-week basis, for a maximum of two weeks. If a stable baseline has not been established by the fourth week, the participant will exit the study and be provided with information about managing distress and accessing further support.

Intervention (Sessions will be audio recorded):

Treatment planning Participants will receive a single face-to-face session at their home, lasting at least one hour up to a maximum of two hours.

Psychoeducation and behavioural activation Participants will receive a single psychoeducation session, followed by three, fortnightly, behavioural activation sessions. In addition, participants will be offered an optional support session for troubleshooting. Sessions will last up to one hour and contact will be made using internet video software.

Treatment evaluation Participants will receive a review session lasting up to one hour, contact will be made using internet video software.

Post-intervention Participants will be contacted by a fellow Trainee Clinical Psychologist to take part in a 30-minute, one-to-one, audio recorded phone interview.

Follow up (Optional) Two months following the treatment evaluation session participants will complete the follow up measures.

Intervention sessions will be audio recorded and then evaluated by an independent researcher from within the sponsors' institution, such as an MSc student. Fidelity will be investigated using a set framework, to investigate alliance, and content delivery adherence. Should participant decline sessions being audio-recorded, fidelity will be checked via session notes.

Data analysis:

Visual analysis will be used to analyse data collected during the intervention. The analysis identifies any phase-related changes in process and outcome variables. The analysis will provide a visual representation of the covariation between process and outcome measures, to explore whether/how the intervention has a positive impact on mood, fatigue, and quality of life. Additionally, visual analysis will be supplemented with use of reliable and clinically significant change indices, to provide quantitative decision criteria for identifying the statistical robustness and practical importance of any visually-apparent shifts over time. A framework analysis will be used to analysis the responses to the change interview.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Secondary Progressive Multiple Sclerosis
* Must speak English
* Must have capacity to give consent
* Must have a telephone
* Must have access to the internet
* Must be able to use a computer
* Must score ≥ 8 on the Hospital Anxiety and Depression Scale - depression subscale

Exclusion Criteria:

• Receiving psychological therapy for a pre-existing mood problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in depression: Hospital Anxiety and Depression Scale; Zigmond & Snaith, 1983 | Screening, Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12
  Measures changes to anxiety and depression over the last one week. The questionnaire is comprised of two scales (anxiety and depression). Each scale has 7 questions, asking participants to rate between 0-3. The questions for each scale are totalled to produce an overall score between 0-21. Higher scores indicate increased severity of anxiety or depression.

SECONDARY OUTCOMES:
Changes to fatigue: Modified Fatigue Impact Scale; Vickrey et al., 1995 | Baseline, Week 6, Week 12
  Measures changes to fatigue. The modified fatigue impact scale is a modified form of the Fatigue Impact Scale (Fisk et al, 1994b) based on items derived from interviews with Multiple Sclerosis patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. Assess the effects of fatigue on quality of life in patients with chronic diseases. Total number of questions 5, asking participants to reflect over the last 4 weeks. The modified fatigue impact scale total score consists of the sum of the raw scores on these 5 items, and thus, can range from 0-20. Higher scores indicate a greater impact of fatigue on a patient's activities.
Changes to quality of life: Health Status Questionnaire Short form version 2. SF-12v2; Ware, Kosinski, & Keller, 1996 | Baseline, Week 6, Week 12
  Measures changes to quality of life. Addresses health concepts from the patient's perspective over 8 domains. The survey uses norm-based scoring
Changes in behaviour associated with depression: The Behavioural Activation for Depression Scale Short Form | Day 1, day 3, day 5, day 7, day 9, day 11, day 13, day 15, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12
  Measures changes in behaviours that underlie depression. Track weekly changes in behaviours that underlie depression and that are specifically targeted for change by Behavioural Activation. Asks 9 questions using a 0-6 scale, comprised of 3 subscales. To score, items from all scales other than the Activation scale are reverse-coded and then all items are summed. To score the subscales, no items are reverse-coded. This process allows high scores on the total scale and the subscales to be represented by the scale and subscale names. In other words, for the total scale, higher scores represent increased activation, while for the Social Impairment subscale, higher scores represent increased social impairment.

OTHER OUTCOMES:
Changes in depression during baseline phase: The Patient Health Questionnaire 2; Kroenke, Spitzer, & Williams, 2003 | Day 1, day 3, day 5, day 7, day 9, day 11, day 13, day 15
  Measures changes to depression. The Patient Health Questionnaire 2 (PHQ2; Kroenke, Spitzer, & Williams, 2003) a two-item questionnaire will be administered every-other-day, during the baseline phase (up to 4 weeks), to establish a baseline for the primary outcome variable of interest (depression). As no higher frequency measure exists questions will be adapted to ask 'over the last two days.' To overcome the impact of adapting the measure, outcome measures such as the Hospital Anxiety and Depression Scale, will be used on a weekly basis.
Changes to valued living: The Engaged Living Scale; Trompetter et al., 2013 | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12
  Measures alignment to values. The scale will be used to identify alignment to values, this will allow us to understand the impact of values-based action. The scale is comprised of 16 items using a 5-point Likert scale. The scale has 2 subscales, Valued Living (10 items) and Life Fulfillment (6 items). Higher scores indicate participants are more aligned to their values.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Moghaddam, PhD, Principal Investigator — University of Lincoln
Locations (1):
- Nottingham University Hospitals - Queens Medical Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No